CLINICAL TRIAL: NCT05006781
Title: The Dose Finding Study of Sodium Benzoate Added to tDCS for the Treatment of Early-phase Alzheimer's Disease
Brief Title: The Dose Finding Study of DAOIB Added to tDCS for AD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was suspended due to the budget issue
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202002208A0
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Transcranial Direct Current Stimulation; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS+Dose A (Experimental): Drug: DAOIB at dose A The DAOIB dose will be fixed during the 24 weeks duration. Device: tDCS tDCS
  Interventions: Drug: DAOIB
- tDCS+Dose B (Experimental): Drug: DAOIB at dose B The DAOIB dose will be fixed during the 24 weeks duration. Device: tDCS tDCS
  Interventions: Drug: DAOIB
- tDCS+Dose C (Experimental): Drug: DAOIB at dose C The DAOIB dose will be fixed during the 24 weeks duration. Device: tDCS tDCS
  Interventions: Drug: DAOIB
- tDCS+placebo (Placebo Comparator): Drug: Placebo Placebo Device: tDCS tDCS
  Interventions: Drug: DAOIB

INTERVENTIONS:
Drug: DAOIB — The DAOIB dose in each group will be fixed during the 24 weeks duration

SUMMARY:
This is a 26-week randomized, double-blind, placebo-controlled trial. We will enroll patients with aMCI or mild AD. All patients will receive 2 weeks of tDCS (5 sessions per week, 10 sessions in total) during the first 2 weeks of the study, and will also be allocated randomly to either of 4 treatment groups for 24 weeks: (1) Dose A group; (2) Dose B group; (3) Dose C group; (4) placebo group. We will assess the patients every 8 weeks during the treatment period (weeks 0, 10, 18, and 26). We hypothesize that augmentation with certain dose of DAOIB will yield better effect than tDCS alone in improving the cognitive function, global functioning and quality of life in patients with aMCI or mild AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease or mild cognitive impairment
* MMSE between 10-26
* CDR 1 or 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 10, 18 and 26 | week 0, 10, 18, 26
  Alzheimer's disease assessment scale-cognitive subscale scores range from 0 (best) to 70 (worst)

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 10, 18 and 26 | week 10, 18, 26
  Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 10, 18 and 26
Change from baseline in Mini-Mental Status examination score at week 10, 18 and 26 | week 0, 10, 18, 26
  Change from baseline in Mini-Mental Status examination score at week 10, 18 and 26
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 10, 18 and 26 | week 0, 10, 18, 26
  The assessment appears to be a suitable instrument for evaluating activities of daily living in early-phase dementia. Its scores range from 0 (worst) to 78 (best)
Change from baseline in Quality of life score at week 10, 18 and 26 | week 0, 10, 18, 26
  Quality of life will be assessed by Medical Outcomes Study Short-Form-36 (SF-36). The SF-36 consists of eight sections: (1) vitality, (2) physical functioning, (3) bodily pain, (4) general health perceptions, (5) physical role functioning, (6) emotional role functioning, (7) social role functioning, and (8) mental health.
Change from baseline in the composite score of a battery of additional cognitive tests at week 26 | week 0, 26
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (Wechsler Memory Scale, Spatial Span), verbal/nonverbal learning and memory tests (Wechsler Memory Scale, Word Listing).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No